

# Rib fracture pain management at a London Major Trauma Centre:

A retrospective comparison of Erector Spinae Plane Blocks, Serratus Anterior Plane Blocks and Thoracic Epidurals

# A retrospective review of rib fracture management at a London Major Trauma Centre comparing Erector Spinae Plane Blocks, Serratus Anterior Plane Blocks and Epidurals V3 06/09/2020

Main Sponsor: Imperial College Healthcare NHS Trust

Ruth Nicholson, Head of Research Governance & Integrity

Imperial College London

Room 215, Level 2, Medical School Building Norfolk Place, St Mary's Hospital Campus

London, W2 1PG

Funders: N/A

Study coordination centre: St Mary's Hospital, Paddington

IRAS ID: 276933



# **Study Management Group**

Chief Investigator: Dr Boyne Bellew

St Mary's Hospital, Paddington Co-investigators: Dr Alex Wickham, Dr Sabena

Qureshi, Dr Claire Broe, Dr Liang Lee, Dr. Andrew Smallbones

Charing Cross Hospital Co-investigators:

Dr Richard Doyle

Statistician: Mr. Roger A'Hern

# **Study Coordination Centre**

For general queries, supply of study documentation, and collection of data, please contact:

Study Coordinator: Dr Boyne Bellew

Address: Department of Anaesthesia & Critical Care,

St Mary's Hospital, Paddington

Anaesthesia / Critical Care / Theatres, Specialist Services - CPG 3

4th Floor, QEQM Building, St Mary's Hospital, Praed Street,

London W2 1NY

# **Clinical Queries**

Clinical queries should be directed to Dr Boyne Bellew who will direct the query to the appropriate person: <a href="mailto:boyne.bellew@nhs.net">boyne.bellew@nhs.net</a>

# **Sponsor**

Imperial College Healthcare NHS Trust is the main research Sponsor for this study. For further information regarding the sponsorship conditions, please contact the Head of Regulatory Compliance at: <a href="mailto:ruth.nicholson@nhs.net">ruth.nicholson@nhs.net</a>

# **Funder**

No funding

This protocol describes the retrospective review of rib fracture pain management at a major trauma centre. Every care was taken in its drafting, but corrections or



amendments may be necessary. These will be circulated to investigators in the study.

This study will adhere to the principles outlined in the Data Protection Act 2018 and General Data Protection Regulations (Europe) and other regulatory requirements as appropriate.

# **Glossary of Abbreviations**

| TARN | Trauma Audit & Research Network |
|------|-----------------------------------|
| ESPB | <b>Erector Spinae Plane Block</b> |
| SAPB | Serratus Anterior Plane Block |
| MTC | Major Trauma Centre |
| ICU | Intensive Care Unit |
| TEA | Thoracic Epidural Analgesia |
| NIV | Non-Invasive Ventilation |

Keywords: Trauma, rib, fracture, analgesia



# **Study Summary**

| Title | Rib fracture pain management at a London Major Trauma |
|---|---|
| | Centre, a retrospective comparison of Erector Spinae Plane |
| | Blocks, Serratus Anterior Plane Blocks and Thoracic Epidurals |
| Design | Single centre retrospective cohort study |
| Aims | To determine whether novel fascial plane blocks, i.e. SAPB |
| | and ESPB, are safe and effective in patients with rib fractures. |
| Outcome Measures | What are the effects of novel regional anaesthesia blocks on: |
| | - Proportion of patients with a reduction in pain |
| | - Pain scores |
| | - Opioid use |
| | - Nausea & vomiting |
| | -Lung complications due to pain |
| | -ICU admission for respiratory complications, |
| | - Use of NIV/invasive ventilation |
| | Block related complications |
| Population | Males and Females |
| Eligibility | Patients aged over 18 with rib fractures |
| Duration | Retrospective review of 5 year period of outcome data |



# Contents

| 1. Introduction | _ |
|---|---|
| 1.1 Background | |
| 1.2 Study Rationale | б |
| 2. Study Objectives | 7 |
| 2.1 Primary Objective | 7 |
| 2.2 Secondary Objectives | 7 |
| 3. Study Design | 7 |
| 4. Study Outcome Measures | 7 |
| 5. Regulatory Issues | 10 |
| 5.1 Ethics approval | 12 |
| 5.2 Consent | 12 |
| 5.3 Confidentiality | 12 |
| 5.4 Indeminity | 11 |
| 5.5 Sponsor | 12 |
| 5.6 Funding | |
| 5.7 Audits | 13 |
| 6. Study Management | 13 |
| 7. Publication Policy | 13 |
| 8. REFERENCES | 14 |
| Appendix A. Imperial NHS Acute Rib Fracture Pathway | 15-32 |



# 1. Introduction

# 1.1 Background

Rib fractures are commonly seen in Trauma Centres around the world, making up two thirds of all chest trauma admissions<sup>1</sup>. In the United Kingdom, 15,000 patients attend hospital with rib fractures annually according to Trauma Audit and Research Network figures. More than a third of these cases develop either short term and or long-term complications, including pneumonia, respiratory failure and chronic pain<sup>2</sup>. Complications typically arise due to poor pain relief in the acute setting.

Pain from rib fractures restricts chest wall movement leading to hypoventilation and impaired coughing ability, which leads to sputum retention and mucus plugging. The injured lung tissue under the fractures also has impaired gas exchange and may contain blood. This causes shunting of blood, ventilation perfusion mismatch, and reduced compliance<sup>3</sup>. These combine to cause atelectasis and increase patients' predisposition to pneumonia. Pneumonia affects up to 30% of patients, with or without sepsis, causing further respiratory compromise. The combination of hypoventilation, atelectasis and/or lobar collapse and impaired gas exchange results in hypoxaemia, respiratory failure and, in some cases, a need for mechanical ventilation. These complications typically develop over 48 – 72 hours following injury<sup>4-7</sup>. The provision of adequate analgesia is widely viewed as a key priority in managing rib injury patients to facilitate improved respiratory effort and enable chest physiotherapy for rehabilitation after rib fractures.

# 1.2 Study Rationale

Thoracic epidural analgesia (TEA) is widely considered to be the current gold standard treatment for rib fracture pain and is used in the Imperial invasive treatment pathway for rib fractures<sup>-1,7</sup> However, TEA are often contraindicated due to other injuries or the use of anticoagulant medications, which also contraindicates other invasive nerve block techniques e.g. paravertebral catheters. A number of case reports have reported the safe use of alternative techniques such as SAPBs and ESPBs<sup>8</sup> and the anaesthesia community has taken them up widely based on this relatively limited evidence. In view of this, Womack et al recently published a large retrospective review examining the safety and efficacy of ultrasound guided paravertebral catheter analgesia techniques in rib fracture management along with small numbers of ESPBs<sup>9</sup>. However, this data did not report the analgesic efficacy, patient reported pain relief or respiratory complications. We wish to advance this body of evidence by reviewing our larger data set concerning the use of TEA and alternative regional techniques such as ESPB



and SAPB. This comprehensive review will benefit patients by documenting the efficacy and safety of these techniques for clinicians managing rib fracture patients.

# 2. Study Objectives

# 2.1 Primary Objective

Our primary objective is to examine whether novel fascial plane blocks, e.g. SAPB and ESPB, are effective pain relief modalities in patients with rib fractures - the proportion of patients with a reduction in pain.

# 2.2 Secondary Objectives

We will review the safety profile and complications of TEA and alternative analgesic techniques such as ESPB and SAPB used for rib fracture management in our trauma centre. In particular, we will examine the effects of regional anaesthesia techniques on:

- 1) Opioid use
- 2) Nausea & vomiting
- 3) Respiratory complications
- 4) Intubation & non-invasive ventilation (NIV)
- 5) ICU admission for respiratory complications

We will assess the duration of use and complication profile of regional anaesthetic techniques, including infection, analyseic failure and damage to other structures during insertion e.g. the lung.

# 3. Study Design

# 3.1 Design & Purpose

A single centre retrospective anonymised data study of a 5 year cohort of rib injury patients managed in a major trauma centre within the Imperial College Healthcare Trust.

# 3.2 Data Collection & Methods

Records will be identified by searching the Trauma Audit and Research Network (TARN) database, a routinely collected database of all patients admitted with traumatic injury within the Imperial College Healthcare Trust. This will be collected by the ICHT TARN co-ordinator. The TARN database provides basic demographic and injury data including hospital number. We will use this information to identify the cohort of patients who were triaged to the Imperial College Healthcare Trust invasive rib fracture care pathway.



Individual patient data will then be obtained from the electronic health record (Cerner) using the patient's hospital number. The data will be pseudo-anonymised and will be collected by members of the study team, all of whom are NIHR Good Clinical Practice trained members of the direct care team. Data will be reviewed and stored on password protected NHS desktop computers in a folder only accessible to members of the study team. Any hard copies of patient data will be stored in a locked filing cabinet within a secure NHS office in St. Mary's Hospital. The study will be conducted from 30/09/2020 until the 31/01/2021. We plan to review rib injured patient's electronic notes that have received these interventions from January 2016 until December 2019 and categorise the information for analysis as set out in study outcomes. Our sample size is estimated at 1200 participants, as per the TARN coordinator. This information will allow us to assess the safety and efficacy of these alternative techniques as compared to TEA.

#### 3.3 Inclusion Criteria

- Patients aged > 18 years of age presenting with traumatic rib fractures in a major trauma centre over the past 5 years
- Meet the criteria for the Imperial College Healthcare NHS Trust 'Invasive rib fracture management pathway' (see Appendix A)

# 3.4 Exclusion Criteria

- Under 18 years old
- Prisoners
- Pregnant
- Private patients
- Meet the criteria for the Imperial College Healthcare NHS Trust 'Non-invasive rib fracture management pathway' (see Appendix A)

# 3.5 Data Analysis

ESP Block (N=~40): The primary hypothesis is that the proportion of patients showing lower pain scores 48-72 hours relative to pain scores at baseline is 70% (approximately 2 out of 3) or more. A rate of 50% or less (1 in 2) would be considered unsatisfactory. With 40 patients it is possible to achieve 80% power at the 5% significance level to distinguish between these two scenarios. The probability that 26 or more of the 40 patients have lower 48-72 hour scores if the true rate is 70% is 81%, if the true rate is 50% there is a 4% chance this will occur. The lower one-sided 95% confidence limit will be presented for the proportion of patients showing lower pain scores at 48-72 hours relative to pain scores at baseline, this estimate will provide a lower limit for the success rate.

SAP Block (N=~35): Similar considerations to those ESPB apply, but in this case the true proportion showing lower pain scores at 48-72 hours would need to be 75% or more to confidently show that the true rate is greater than 50%. For example, the probability that 23 or



more of the 35 patients have lower 48-72 hour scores (if the true rate is 75%) is 92%, if the true rate is 50% there is a 4.5% chance this will occur.

TEA (N=~250)

The large number of subjects in this group means that the aim of distinguishing 70% versus 50% success rates can be confidently achieved, with a power of more than 99% at the 5% significance level.

Generally, for binary endpoints, 95% confidence intervals for the proportions of at most +/- 17% can be estimated for SAP Block subjects, +/- 16% for ESPB subjects and +/- 7% for TEA subjects.

# 4. Study Outcome Measures

# **4.1 Primary Outcome Measure**

We aim to review pain scores as recorded by clinical staff over 72 hours to assess pain relief efficacy, A verbal rating scale classifying pain as mild, moderate or severe is used at Imperial Data from the acute pain round records will also provide details regarding breathing comfort levels of the patient, coughing ability and deep inspiratory effort. These are recorded as yes/no answers and we will assess the proportion of patients showing a reduction in pain scores.

# **4.2 Secondary Outcome Measures**

### 4.2.1 Indication for the nerve block

All patients with rib fractures who met the criteria for the invasive rib fracture care pathway as set out in Appendix A. The diagram below describes the main criteria for allocation to the invasive or non-invasive pathway for rib fracture pain management.



### Risk factors for morbidity

Pulmonary contusion Current smoker Cardiovascular disease Frailty Presence of ≥2 distant injuries Obesity & OSA

# Early review for surgical rib fixation

Flail chest Chest wall deformity
≥3 displaced rib fractures CXR: ≥25% lung volume loss
≥65 years old NIV/ ventilator dependent

# Start on appropriate arm of pathway



# **S**

# Battle score 0 - 15



# Battle Score ≥16

# Non Invasive

If score 0 – 10: consider CDU if meets criteria or discharge if appropriate

If score 11 – 15 or other risk factors for morbidity present: consider more advanced analgesia & escalation to invasive pathway

# Invasive

If score  $\geq$ 30: consider early liaison with critical care team

# 4.2.2 A marker of injury severity e.g. Battle score

Table 4 Risk factor scores as transformed from the regression coefficients

| | Regression coefficient | Risk score |
|------------------------------|------------------------|----------------|
| Age | 0.0162 | 1ª |
| Number of rib fractures | 0.418 | 3 <sup>b</sup> |
| Chronic lung disease | 0.789 | 5 |
| Pre-injury anticoagulant use | 0.637 | 4 |
| Oxygen saturation levels | -0.0651 | 2 <sup>c</sup> |
| 3 | b | |

<sup>&</sup>lt;sup>a</sup>Per additional 10-year increase starting at 10 years of age; <sup>b</sup>per additional rib fracture; <sup>c</sup>per 5% decrease in oxygen saturations starting at 94%.

Table 5 Final risk scores and corresponding probability of developing complications

| Final risk score | Probability mean ± SD |
|------------------|-----------------------|
| 0 to 10 | 13% ± 6 |
| 11 to 15 | 29% ± 8 |
| 16 to 20 | 52% ± 8 |
| 21 to 25 | 70% ± 6 |
| 26 to 30 | 80% ± 6 |
| 31+ | 88% ± 7 |

Table 3. Rib fracture risk score adapted from Battle et al<sup>2</sup>

| Variable | Score | Example |
|---|---|---|
| Age | +1 per additional 10-year increase starting at 10 years of age | 4 |
| Number of rib fractures | +3 per rib fractured | 15 |
| Chronic lung disease | +5 if present | 5 |
| Pre-injury anti-coagulant use | +4 | 0 |
| Peripheral oxygen saturation levels (SpO <sub>2</sub> ) | +2 per 5% decrease SpO <sub>2</sub> starting at 94% at time of assessment | 2 |
| Total | | 26 |

# 4.2.3 Morphine based products/other analgesic medications used



Data regarding type of opiate use, mode of delivery, dosage requirement in 24 hours and complications associated with opiates such as constipation, delirium and respiratory depression.

# 4.2.4 Nausea & vomiting

The incidence of nausea and vomiting pre-chest wall block and in the 72 hours post block will be recorded with the number of episodes and number of anti-emetic medications required to treat.

# 4.2.5 Lung complications as a result of pain

- 1) Lower Respiratory Tract Infection (LRTI): for this study is defined as patients showing clinical features of chest infection including pyrexia (temperature >37.5°C), an increase in oxygen requirements from baseline, radiological evidence of chest infection or antimicrobial treatment of an LRTI started by the treating team.
- 2) Empyema/Parapneumonic effusions: defined as radiological evidence of fluid collections within the pleural space and therapeutic interventions required for treatment e.g. aspiration and drainage.

#### 4.2.6 Intensive care admission

- ICU admission for respiratory complications
- -Number of patients requiring intubation and ventilation
- Number of days of mechanical ventilation
- -Length of ICU stay

# 4.2.7 Other nerve block complications

- 1) Block failure: defined as persistent moderate to severe pain following insertion of TEA, ESPB or SAPB catheters in spite of adequate dosing of analgesia at any time after initial placement.
- 2) Number of catheter resiting events
- 3) Number of catheter top-ups required within a 24 hour period
- 4) Regional anaesthetic catheter associated infection
- 5) Pneumothorax secondary to regional anaesthesia technique



# 5. Regulatory Issues

# 5.1 Ethics approval

The Chief Investigator has obtained approval from the Health Research Authority. The study must also receive confirmation of capacity and capability from each participating NHS Trust before starting the study. The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Helsinki 1964 and later revisions

# 5.2 Consent

This is a retrospective case notes review study. This data is collected as routine care and for the TARN database. As the study only involves retrospective data collection at a single time point that will not impact clinical care, obtaining informed consent is not necessary. The only personal identifiable information we intend to collect is the hospital number, which is pseudonomyised. Each patient has a unique number according to their order within the data excel spreadsheet and the link to these will be recorded and stored on a password protected disc stored on password protected NHS Trust computers accessible only by members of the study team.

# 5.3 Confidentiality

This is a retrospective pseudo-anonymized data collection study of available clinical data so no consent is needed. Data will be extracted and reviewed by members of direct care team who are also members of the research team. Only anonymized data will be analysed and published. All identifiable information will be securely held in NHS Trust computers and there will be held in strict compliance to NHS Data Protection and Confidentiality regulation. The Chief Investigator will preserve the confidentiality of participants taking part in the study and is registered under the Data Protection Act. Data and all appropriate documentation will be stored for 5 years after the completion of the study, including the follow-up period. If data is missing this will be stated and not included in the final data analysis. i

We will employ the use of passwords to restrict access to electronic documents and store hard copies of study documents in a locked cabinet in secured location within the anaesthetic department at St Mary's Hospital. The data will only be accessible by the research team involved in the project. Only pooled population data will be used in outputs.

# 5.4 Indemnity

Imperial College Healthcare NHS Trust holds standard NHS Hospital Indemnity and insurance cover with NHS Resolution for NHS Trusts in England, which apply to this study



# 5.5 Sponsor

Imperial College Healthcare NHS Trust will act as the main Sponsor for this study. Delegated responsibilities will be assigned to the NHS trusts taking part in this study.

# 5.6 Funding

No funding is required for this study.

# 5.7 Audits

The Joint Research Compliance Office, Imperial College London Imperial College Healthcare NHS Trust may audit the study.

# 6. Study Management

The day-to-day management of the study will be co-ordinated through Dr Boyne Bellew.

# 7. Publication Policy

The study results will be presented at specialty conferences and published in a peer reviewed anaesthetic journal. No patient identifiable information will be included.



# 8. REFERENCES

- 1. Simon, B. J. et al. (2005) 'Pain Management Guidelines for Blunt Thoracic Trauma', The Journal of Trauma: Injury, Infection, and Critical Care, pp. 1256–1267. doi: 10.1097/01.ta.0000178063.77946.f5.
- 2. The Trauma Audit and Research Network. Performance comparison: northern. 2018. www.tarn.ac.uk/Content.aspx? ca=15&c = 3468 (accessed 01/06/2018).
- 3. Ahn, Y. et al. (2013) 'Pain-associated Respiratory Failure in Chest Trauma', Anesthesiology. The American Society of Anesthesiologists, 118(3), pp. 701–708. doi: 10.1097/ALN.0b013e318283996b.
- 4. Barnea, Y. et al. (2002) 'Isolated rib fractures in elderly patients: mortality and morbidity.', Canadian journal of surgery. Journal canadien de chirurgie. Canadian Medical Association, 45(1), pp. 43–6. Available at: http://www.ncbi.nlm.nih.gov/pubmed/11837920 (Accessed: 4 June 2019).
- 5. Jones, K. M., Reed, R. L. and Luchette, F. A. (2011) 'The ribs or not the ribs: which influences mortality?', The American Journal of Surgery. Elsevier, 202(5), pp. 598–604. doi: 10.1016/J.AMJSURG.2010.09.029.
- 6. May, L., Hillermann, C. and Patil, S. (2016) 'Rib fracture management', BJA Education. Narnia, 16(1), pp. 26–32. doi: 10.1093/bjaceaccp/mkv011.
- 7. Witt CE, Bulger EM (2017) 'Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol' Trauma Surgery & Acute Care Open 2017;2:e000064. doi: 10.1136/tsaco-2016-000064
- 8. Adhikary, S. D. et al. (2019) 'The effect of erector spinae plane block on respiratory and analgesic outcomes in multiple rib fractures: a retrospective cohort study', Anaesthesia. John Wiley & Sons, Ltd (10.1111), 74(5), pp. 585–593. doi: 10.1111/anae.14579.
- 9. Womack, J at al. (2019) "Safety, complications and clinical outcome after ultrasound-guided paravertebral catheter insertion for rib fracture analgesia: a single-centre retrospective observational study; Anaesthesia 2019, 74, 594–601, doi:10.1111/anae.14580



# Appendix A. Imperial NHS Acute Rib Fracture Pathway

# 1) **SUMMARY**

This revised guideline provides a framework for the assessment and management of adult patients with rib fractures at Imperial College Healthcare NHS Trust. The guideline has been updated to take account of new evidence in patient risk assessment, analgesic management strategies and physiotherapy techniques. Additionally, criteria for accepting referrals for tertiary level care of rib fractures are provided.

# 2) INTRODUCTION

# 2.1 Incidence

Blunt chest-wall trauma accounts for 10-15% of all trauma admissions to Emergency Departments (EDs) globally<sup>1,2</sup>. Rib fractures may complicate up to two thirds of these injuries<sup>2</sup>. North West London Trauma Network treats approximately 450 patients with rib fractures per year, of whom approximately two thirds receive tertiary care at St Mary's.

# 2.2 Importance

Rib fractures are markers of severe injury and are associated with significant morbidity and mortality. Patients with these injuries are at greater risk of complications and poor outcomes<sup>2-4</sup>. Associated injuries occur in 94% of patients, typically concomitant thoracic trauma, but also injuries to the head, abdomen and limbs<sup>3</sup>. Mortality associated with rib fractures is hard to calculate, as death often happens indirectly, however it has been estimated as between 10–13%<sup>3,4</sup>, with one article reporting up to 30%<sup>5</sup>. Common immediate thoracic rib include seguelae fractures pneumothorax. haemothorax. haemopneumothorax, pneumatocoele, pulmonary contusions. Solid organs, such as the liver, kidneys and spleen, may also sustain lacerations from broken ribs<sup>1</sup>.

Pain is the most common symptom from rib fractures and a key component in pulmonary complications. Pain restricts tidal volume, leading to hypoventilation, and impairs coughing ability, leading to sputum retention; these combine to cause atelectasis and predispose to pneumonia. Additionally, injured lung tissue underlying the fractures has impaired ability to exchange gasses (leading to shunt and VQ mismatch) and reduced compliance. Compensatory increases in respiratory rate may increase oxygen consumption. Pneumonia occurs in up to 30% of cases, with or without sepsis, causing further respiratory compromise. The combination of hypoventilation, atelectasis and/or lobar collapse and impaired gas exchange results in hypoxaemia, respiratory failure and, in some cases, a need for mechanical ventilation. Respiratory complications typically develop at 48 – 72 hours post injury. Other respiratory complications include pulmonary embolus, pulmonary effusions, empyema and acute respiratory distress syndrome (ARDS)<sup>1-6</sup>.

Patients with rib fractures often require hospital admission, and in more significant injuries, to level 2 or 3 care. The associated incremental costs have not been fully evaluated, but can be considered in terms of length of inpatient stay, 'ICU bed days' and 'ventilator days' and are likely to be significant. Studies evaluating longer term outcomes have demonstrated high rates of chronic disability and chronic pain<sup>3,6,7,10</sup>. The severity of acute pain predicts chronic pain whilst disability is predicted by acute pain intensity and the presence of bilateral



fractures<sup>10</sup>. Elderly patients (aged 65 years or older), have been consistently shown to have worse outcomes, higher complication rates and greater mortality after rib fractures than younger patients<sup>3,7</sup>.



# 3) **DEFINITIONS**

- Rib fracture: a break in a bone making up the rib cage.
- Flail chest: at least 2 fractures per rib in at least 2 adjacent ribs are needed to produce a flail segment. Flail segments cause paradoxical inspiratory movements, compromise breathing and may be life threatening.
- Verbal Rating Scale: a method for assessing pain on an alphanumeric scale. ICHNHST recommends mild, moderate and severe, whilst in the ED the numerical scale 0-10 is used.
- Thoracic Epidural (TE): a fine bore catheter placed into the thoracic epidural space which is used to give analgesic drugs.
- Paravertebral block (PVB): regional anaesthetic technique providing analgesia to a segment of one hemithorax.
- Patient Controlled Analgesia (PCA): a method of allowing a patient to administer their own analgesia intravenously, usually opioid based.
- Non-invasive ventilation (NIV): facial Continuous Positive Airways Pressure (CPAP) or Bi-level Positive Airways Pressure (BIPAP) ventilation
- Morphine Immediate Release (IR): a morphine immediate release preparation (available as a liquid commonly known as Oramorph and tablets)
- Oxycodone Immediate Release (IR): a oxycodone immediate release preparation (available as a liquid and capsules)

# 4) SCOPE

These guidelines are for all staff involved in the care of adult trauma patients with rib fractures but are of particular relevance to those working in the Emergency Department, Theatres, Anaesthesia, Major Trauma Ward and other wards receiving trauma patients. They may also be adopted more widely within the North West London Trauma Network.



# **FULL GUIDELINE**

The use of multidisciplinary bundled care pathways is associated with improved outcomes in patients with rib fractures/ blunt chest injury<sup>3,24</sup>.

# 4.1 Identifying the high-risk patient

Multiple risk factors have been identified for poor outcomes in rib fractures, but the variables can be simply classified into anatomical, physiological and other categories, see table 1.

Many scoring systems are available to predict the risk of complications after blunt chest trauma, all of which combine different variables from table 1. These include the AIS<sub>chest</sub>, Pulmonary Contusion score (PCS), Wagner-score, the Thoracic Trauma Severity score (TTS), the Chest Trauma Score (CTS), RibScore and Easter's Rib Fracture Score. Battle *et al* recently used robust methodology to develop an up to date risk prediction tool that is based on a UK population<sup>2</sup>. The risk of developing complications increases with an increasing score, *see table 2* for details.

Table 1: risk factors for morbidity after rib fractures<sup>1-8</sup>

| Anatomical | Physiological | Other |
|---|---|---|
| <ul> <li>Number of ribs fractured</li> <li>Presence of flail segment</li> <li>Bilateral rib fractures</li> <li>First rib fractured</li> <li>Degree of fracture displacement</li> <li>Fractures in the anterior, lateral and posterior regions</li> <li>Presence of pulmonary contusions</li> <li>Presence of ≥2 distant injuries</li> </ul> | <ul> <li>Reduced physiological reserve: <ul> <li>Increasing age</li> <li>Premorbid respiratory disease</li> <li>Smoking</li> <li>Overweight or obese (BMI &gt;25)</li> <li>Obstructive sleep apnoea</li> <li>Premorbid cardiovascular disease</li> <li>Premorbid diabetes</li> </ul> </li> <li>Reduced SpO₂ at presentation</li> <li>Reduced vital capacity (VC)</li> <li>Post injury pneumonia</li> </ul> | <ul> <li>Premorbid use of anticoagulants</li> <li>Treated in low volume centres</li> <li>Treated outwith a pathway</li> </ul> |

Table 2. Rib fracture risk score and risk of complications from Battle et al<sup>2</sup>

| Final risk score | Probability mean $\pm$ SD |
|------------------|---------------------------|
| 0 to 10 | 13% ± 6 |
| 11 to 15 | 29% ± 8 |
| 16 to 20 | 52% ± 8 |
| 21 to 25 | 70% ± 6 |
| 26 to 30 | $80\% \pm 6$ |
| 31+ | 88% ± 7 |

Battle's tool has been incorporated into the pathway to guide enrolment into the non-invasive (simple analgesia) or invasive (incorporating advanced analgesic techniques) pathway with a cut off point of 15. An example case of a 58 year old man with COPD who has sustained 5 rib fractures and has oxygen saturations of 94% is provided in table 3.

Table 3. Rib fracture risk score adapted from Battle et al<sup>2</sup>

Age

+1 per additional 10-year increase starting at 10 years of age



| Number of rib fractures | +3 per rib fractured | 15 |
|---|---|---|
| Chronic lung disease | +5 if present | 5 |
| Pre-injury anti-coagulant use | +4 | 0 |
| Peripheral oxygen saturation levels (SpO <sub>2</sub> ) | +2 per 5% decrease SpO <sub>2</sub> starting at 94% at time of | 2 |
| | assessment | |
| Total | | 26 |

Objective measures of respiratory function, such as peak expiratory flow rate (PEFR), inspiratory volume (ISV) and vital capacity (VC) have been evaluated<sup>8,9</sup>. VC less than 30% of a patients



predicted value predicts pulmonary complications and each 10% increase in VC is associated with a reduced chance of pulmonary complications (odds ratio 0.64)<sup>9</sup>. The risk of complications can be reduced by adhering to the key principles of management: optimal analgesia, respiratory support, early mobilisation and appropriate surgical intervention.

# 4.2 Analgesic options

As pain is a significant contributor to the morbidity arising from rib fractures, optimisation of analgesia is key to preventing complications. There are many options for managing pain from rib fractures including multimodal oral therapy, intravenous analgesia, topical treatments and a variety of regional anaesthetic blocks.

Acute pain should be assessed according to the Imperial College Healthcare NHS Trust Acute Pain Guideline. In particular for rib fracture patients, assess pain at rest and on coughing/ deep inspiration and ask about features of neuropathic pain for example tingling, burning and electric shock like sensations. Multimodal oral analgesia should be started on admission and include regular paracetamol, ibuprofen and opioids. Morphine should be prescribed both regularly and for breakthrough (PRN).

In patients aged 65 years or older, ibuprofen should be omitted and the regular opioid changed to oxycodone, which has a better pharmacokinetic profile for elderly patients. In patients with renal impairment, defined as eGFR <30mls/min, ibuprofen should be omitted and the oxycodone dose reduced. All patients should receive adjunctive treatments for opioid analgesia including laxatives and anti-emetics. See figure 1 for details.

Opioids may be administered via a patient controlled analgesia (PCA) device if the pain requires more frequent opioid dosing than the standard prescription allows. Patients with features of neuropathic pain such as burning, tingling, electric shock like sensations or numbness should be prescribed a gabapentinoid.

Ketamine may be trialled intravenously (up to 10mg) and continued orally or as an infusion, following the Imperial College Healthcare NHS Trust guidelines, in patients with difficult to manage pain. In any patient with pain that is difficult to control using conventional measures, conversion to the invasive pathway should be considered. (Note the use of ketamine in pain management is unlicensed).

All regional anaesthetic techniques for rib fracture analgesia impair impulse transmission at various points along the intercostal nerve. Thoracic Epidural analgesia remains the gold standard analgesic modality. They are the most widely studied mode of analgesia, and their use in rib fractures is endorsed by several systematic reviews and international bodies<sup>1,3,7</sup>. Expertise at St Mary's allows for timely epidural insertion by senior anaesthetists and appropriate management once sited. Despite this, epidurals have a low but significant complication rate<sup>11</sup> and in some patients may be contraindicated (see table 4); there is also an inevitable failure rate and their benefit has been questioned<sup>12</sup>. Thoracic epidurals and blocks should only be inserted, doses titrated and drugs bolused by appropriately trained members of healthcare staff. The first line epidural infusion should be mixed levobupivacaine 0.125% with fentanyl 2micrograms/mL. In patients with rib fractures and other injuries arising from the same incident, a plain 0.125% levobupivacaine epidural infusion can be started in conjunction with an opioid PCA. Commencing and caring for a patient with an epidural infusion should follow the clinical guideline *Epidural Analgesia: Continuous Infusions Clinical Guidelines for Adult Patients*.



# Table 4: Contra-indications to epidural analgesia. Starred items apply to regional blocks

# Contraindications to epidural analgesia

| Absolute | | te Relative | | | 2 |
|---|---|---|---|---|---|
| 1.<br>2.<br>3. | Patient refusal*<br>Spinal cord injury or haematoma<br>Epidural haematoma | | to position patient*<br>atic Brain Injury with | 5. | Coagulopathy: INR >1.4 or platelets <80 x 10 <sup>9</sup> /L* |
| 4. | Thoracic vertebral body fracture at level of insertion | 3. Incomp | rolled Intracranial Pressure<br>plete spinal evaluation | 6. | Active Anticoagulant therapy. AAGBI RAPAC guide.* |
| 5. | Local or generalised sepsis* | 4. Previo | us thoracic spinal surgery | 7. | Extubation not anticipated within 5 days (ICU patients)* |
| 6. | Open wound at site of insertion* | | | | |



Alternatives to epidurals include intercostal, interpleural and paravertebral blocks, but all have significant drawbacks and lack evidence of benefit over epidurals<sup>13</sup>. Newer techniques, including serratus anterior plane and erector spinae plane blocks, have not yet been robustly evaluated<sup>14,15,23</sup> in the rib fracture population but are used in some trauma units and are the subject of much research interest. They may be of use in patients with unilateral injuries, when thoracic epidurals are contraindicated or are not possible to insert.

In addition to trauma specific cautions and contra-indications (see table 4), standard cautions should be applied prior to inserting an epidural or regional anaesthetic block. Invasive monitoring and critical care should be considered in patients with pre-existing comorbid disease that may be affected by an epidural or regional block e.g. stenotic valvular heart lesions.

# **4.3 Ventilation Management**

Rib fractures are commonly associated with underlying pulmonary contusions and pleural injuries such as pneumothorax and haemothorax. These, combined with pain, can lead to respiratory failure.

To prevent complications and ensure a timely recovery, all patients admitted with rib fractures should receive respiratory support titrated to their individual needs. Patients should be managed on wards with nursing staff familiar with the injury. Supplemental oxygen should be prescribed and administered at the lowest concentration required to achieve peripheral oxygen saturations (SpO<sub>2</sub>) of 94-98%, or 88-92% in patients at risk of carbon dioxide retention. If more than 2-4L/min via nasal cannulae is required, administered oxygen should be humidified to loosen secretions. Sodium chloride (NaCL) 0.9% nebulisers may be prescribed as required or regularly to assist expectoration. Salbutamol nebulisers can be prescribed for bronchospasm. Patients should be mobilised where possible and when in bed, be nursed sitting as upright as possible with attention to pressure area care. All rib fracture patients should receive physiotherapy input at least once a day (see below) until respiratory function normalises and mobility restored to baseline.

Advanced respiratory support including Continuous Positive Airways Pressure (CPAP), Non-Invasive Ventilation (NIV) and Nasal high flow oxygen (Optiflow/ Airvo etc) can be considered, in liaison with critical care staff, for patients with anticipated or deteriorating respiratory failure. Decisions regarding which of these treatment modalities is appropriate will be specific to individual patients and determined by the clinical judgement of the attending trauma, anaesthetic and critical care teams. Patients with significant flail segments in particular should be referred early for critical care review regarding advanced respiratory support, even without evidence of respiratory failure, with the goal of maintaining lung volume and effective cough. A proactive approach to Chest X-Rays should be adopted for patients with flail segments; changes such as atelectasis warrant prompt referral to critical care. Preventative ventilatory support is a key strategy that must be adopted.

# 4.4 Physiotherapy

Physiotherapy should be started within 24 hours of admission in all patients to support ventilation and prevent complications. The ability of patients to participate in physiotherapy is dependent on adequate analgesia using non-sedative doses.

All patients should be taught to perform a simple active cycle breathing technique (ACBT), huffing and encouraged to cough. This can be initiated by nursing staff if necessary, for example at weekends and in the evenings. ACBT consists of taking 3-5 deep breaths with an inspiratory hold of 2-3 seconds followed by 3 relaxed breaths. Patients should be asked to complete ACBT hourly when awake. Instructions for patients (adapted from the <u>Association of Chartered Physiotherapists in Respiratory Care leaflet GL-05</u>):

- 1. Please take a long, slow, deep breath in, ideally through your nose.
- 2. Hold your breath for 2-3 seconds.
- 3. Breathe out gently, like a sigh.
- 4. Repeat this technique for 3-5 breaths approximately every hour.



Huffing is a rapid exhalation of air through an open mouth and throat, as if trying to mist up a mirror. It helps to move sputum up the airways from where it can be coughed out. Huffing should be followed by the deep breathing cycle described above.

In patients who are able to mobilise, early and regular mobilisation should be encouraged. Exercise bikes/floor pedal exercisers can be provided to assist patients who are only able to move into a chair. Shoulder exercises should be taught in appropriate patients to prevent movement restrictions post injury which can limit return to work.

# 4.5 Surgery

Surgical fixation and stabilisation of flail chest injuries is associated with reductions in duration of mechanical ventilation, ICU stay, total hospital stay, hospital acquired pneumonia and mortality rates<sup>16-20</sup>. In the long term patients return to work sooner and have a reduced incidence of chronic pain and analgesic dependence<sup>18-22</sup>. Studies have also shown similar beneficial outcomes in patients with multiple rib fractures but without a flail segment<sup>21</sup>. A multidisciplinary approach to patient selection for surgery is essential. The National Institute of Clinical Health and Excellence has approved and issued guidance on surgical fixation of flail chest injuries<sup>22</sup>.

# 4.6 Referral criteria for tertiary care in North West London Trauma Network

Many patients with rib fractures will present to trauma units within the North West London Network. Some may require tertiary level services, however, the majority can receive care and pain relief at their local trauma unit following local rib fracture pain management guidelines.

Indications for referral to St Mary's Major Trauma Centre are detailed below. Acute referrals should be made to the Trauma Team Leader (TTL) on duty via the TTL mobile or bleep 1328 via switchboard. Internal referrals for consideration of rib fixation should be made to the rib fracture team, via e-mail (imperial.ribfracture@nhs.net).

- 1. Rib fractures associated with:
  - a. Significant pneumothorax
  - b. Haemothorax
  - c. Flail segment
  - d. Moderate/significant pulmonary contusions
- 2. Rib fractures in a polytrauma patient.
- 3. Consideration for rib fracture fixation. Indications (adapted from NICE IPG 361)<sup>22</sup> include:
  - a. Clinical evidence of flail chest (visible paradoxical chest movements) associated with respiratory failure
  - b. ≥3 displaced rib fractures not responding to adequate analgesia
  - c. Significant chest wall deformity or ≥25% lung volume loss on CXR
  - d. Bilateral rib fractures
  - e. Non-invasive ventilation/invasive ventilation dependent
  - f. Presence of clavicle or scapular fracture

# 4.7 Placement of patients at St Mary's Hospital

Most patients will be admitted onto the major trauma, orthopaedic or general surgical wards, but some patients can be admitted elsewhere. Patients with thoracic epidurals should be admitted to major trauma ward or the critical care complex.

#### Clinical Decision Unit

Patients with rib fractures can be considered for admission to CDU only if they meet certain criteria:

• Patients 65 years or older: less than or equal to 2 ribfractures.



- Patients aged under 65 years: less than or equal to 3 ribfractures.
- Exclusion criteria for all age groups:
  - Injury includes: flail segment, significant pneumothorax or haemothorax.
  - Pain relief: requires PCA, epidural or block.



Patients with isolated rib fractures, meeting CDU criteria, who are well pre-injury and who have adequate social support can be considered for immediate or early discharge. Such patients should be counselled to seek medical advice if symptoms change or deteriorate.

#### **Intensive Care Unit**

Patients in ICU receiving level 2 care should follow the standard non-invasive or invasive pathway as appropriate. Patients who would benefit from non-invasive ventilation should also be considered for arterial line insertion and regular blood gases to assess respiratory function.

In patients who are receiving level 3 care (i.e. sedated, intubated and ventilated), the following principles should be considered:

# Ventilation:

- Use lung protective ventilation strategies.
- Nurse with the head of the bed elevated to ≥30 degrees if not contraindicated by other injuries.
- Regular subglottic suctioning.

#### Analgesia:

- Assess pain regularly and treat with multimodal analgesic therapy.
- Contact 1201 to arrange for a thoracic epidural:
  - In patients showing signs of impaired respiratory effort e.g. tachypnoea, poor tidal volumes, signs of pain or the patient indicates they are in pain.
  - In the 24 hours prior to planned extubation in patients meeting the invasive pathway criteria.
- Consider referral for rib fixation (and concurrent epidural) if:
  - o Flail chest or paradoxical chest movement during weaning from a ventilator
  - > 6 ribs fractured
  - Bilateral rib fractures
  - Hypoxia and/or hypercarbia under 40% inspired oxygen inhalation
  - o Repeated atelectasis
  - Significant chest wall deformity
  - o Not responding to thoracic epidural and do not require intubation and ventilation otherwise

# 4.8 Discharge

Prior to discharge, patients should be given information, for example the <a href="NHS choices">NHS choices</a> rib injury sheet, to ensure their progress after discharge is optimal. Pain should be adequately controlled such that patients are discharged with weak opioids (as well as other multimodal agents) in the TTO pack. If stronger opioids, e.g. morphine, are still in use, a clear weaning plan should be in place for the GP. Patients should be advised to see their GP if the pain isn't responding to prescribed analgesics or if they develop features of chest infection. Other simple interventions that can be recommended for completion at home include continued use of the active cycle breathing technique, use of ice packs, use of splints when coughing (e.g. a rolled-up towel), encouragement of mobilisation but avoidance of heavy strenuous exercise or work. Patients who have received surgical rib fracture fixation should be followed up in fracture clinic at 6 weeks after discharge.



Figure 1: Overview of Imperial rib fracture pathway

# Rib Fracture Pathway Overview

# 1 Rib fractures confirmed on CXR / CT



# 2 Start multimodal analgesia and adjuncts

| Adult patients |
|---|
| Paracetamol 1g PO/ IV 6 hourly<br>(if weight <50kg dose at 15mg/kg IV) |
| Morphine IR* 10 - 20mg PO 4 hourly<br>+<br>Morphine IR* 5 – 10mg PO 4 hourly PRN |
| Ibuprofen 400mg PO QDS |
| Laxatives: macrogol 1 sachet BD and senna 15mg ON |
| Anti-emetics |

| Patients aged 65yrs or older |
|------------------------------------------------------------------------|
| Paracetamol 1g PO/ IV 6 hourly<br>(if weight <50kg dose at 15mg/kg IV) |
| Oxycodone IR* 2.5 – 5mg PO 4 hourly |
| Oxycodone IR* 2.5 – 5mg PO 4 hourly PRN |
| Avoid NSAIDs |
| Laxatives: macrogol 1 sachet BD and senna 15mg ON |
| Anti-emetics |

| Patients with renal impairment (eGFR <30) |
|------------------------------------------------------------------------|
| Paracetamol 1g PO/ IV 6 hourly<br>(if weight <50kg dose at 15mg/kg IV) |
| Oxycodone IR* 1.25 – 2.5mg PO 4 hourly + |
| Oxycodone IR* 1.25 – 2.5mg PO 4 hourly PRN |
| Avoid NSAIDs |
| Laxatives: macrogol 1 sachet BD and senna<br>15mg ON |
| Anti-emetics |
| *ID - Immediate Delegae |

\*IR = Immediate Release

# Assess Risk (Battle's score)

| Variable<br>_Age | Score<br>. +1 per additional 10-year increase starting at 10 years of age |
|---|---|
| Number of rib fractures | +3 per rib fractured |
| Chronic lung disease | +5 if present |
| Pre-injury anti-coagulant use | +4 |
| Peripheral oxygen saturation levels (SpO <sub>2</sub> ) | +2 per 5% decrease SpO <sub>2</sub> starting at 94% at time of assessment |
| Total | |

# Please document Battle score on Cerner

Consider other risk factors for morbidity and the need for fib fixation:

# Risk factors for morbidity

# Early review for surgical rib fixation

Pulmonary contusionCurrent smokerFlail chestChest wall deformityCardiovascular diseaseFrailty≥3 displaced rib fracturesCXR: ≥25% lung volume lossPresence of ≥2 distant injuriesObesity & OSA≥65 years oldNIV/ ventilator dependent

# 4 Start on appropriate arm of pathway







Battle score 0 – 15



# Non Invasive

If score 0-10: consider CDU if meets criteria or discharge if appropriate

If score 11 – 15 or other risk factors for morbidity present: consider more advanced analysis &

Battle Score ≥16



# **Invasive**

If score  $\geq$ 30: consider early liaison with critical care team



Figure 2: Non-Invasive pathway for rib fracture management

# Non - Invasive Pathway

Nursing care provided by staff familiar with major trauma patients Monitor oxygen saturation (SpO<sub>2</sub>) and Vital Capacity



Encourage to sit upright and mobilise early where possible

Provide supplemental oxygen at the lowest contentration to achieve appropriate SpO<sub>2</sub>

# 3 Confirm analgesia is prescribed and titrate as required

| Adult patients Paracetamol 1g PO/ IV 6 hourly | Patients aged 65yrs or older Paracetamol 1g PO/ IV 6 hourly | Patients with renal impairment (eGFR <30) Paracetamol 1g PO/ IV 6 hourly |
|---|---|---|
| (if weight <50kg dose at 15mg/kg IV) Morphine IR* 10 – 20 PO 4 hourly | Oxycodone IR* 2.5 – 5mg PO 4 hourly | (if weight <50kg dose at 15mg/kg IV) Oxycodone IR* 1.25 – 2.5mg PO 4 hourly |
| + | +<br>Avoid NSAIDs | |
| Morphine IR* 5 – 10mg PO 4 hourly PRN Ibuprofen 400mg PO QDS | Laxatives: macrogol 1 sachet BD and senna 15mg ON Anti-emetics | Oxycodone IR* 1.25 – 2.5mg PO 4 hourly PRN Avoid NSAIDs |

Consider IV opioid PCA: Morphine 1<sup>st</sup> choice, Fentanyl 2<sup>nd</sup> choice (unless renal impairment). Give pregabalin if features of neuropathic pain. Consider PO ketamine after successful IV trial. Contact pain team (bleep 1043) or anaesthetic\_team (bleep 1213) for advice

Active Cycle Breathing Technique including "huffing" hourly when awake Encourage early and regular mobilisation for those able

Pedal exercisers for patients unable to mobilise beyond a chair

# 5 Regular reassessment and titration of therapy



 $SpO_2/PaO_2/Vital$  Capacity reducing  $O_2$  needs increasing

SpO<sub>2</sub>/ PaO<sub>2</sub>/ Vital Capacity improving/ stable
O<sub>2</sub> needs reducing/ stable



Figure 3: invasive pathway for rib fracture management

# Invasive Pathway

Nursing care provided by staff familiar with major trauma patients Monitor oxygen saturation (SpO<sub>2</sub>) and Vital Capacity



As per items 2-4 on the Non-Invasive Pathway



TE is the 1<sup>st</sup> choice block for rib fractures. If there are contraindications, consider a block.

Both should be booked under "Emergency NCEPOD" on Cerner and completed within 6 hours of admission.

#### No contraindications

# **Thoracic Epidural**

Initial bolus of 10 – 15mls levobupivacaine 0.125%

Prescribe mixed bag levobupivacaine 0.125% + 2mcg/ml fentanyl at 15mls/hr + rescue bolus 10mls





TE

Serratus Anterior or Erector Spinae Plane Block Initial bolus of 40mls levobupivacaine 0.125% + 1:400000 adrenaline

Prescribe plain levobupivacaine 0.125% at 15mls/hr + rescue bolus 20mls 4 hourly PRN

# contraindicated





# A Regular reassessment and titration of therapy SpO<sub>2</sub>/ PaO<sub>2</sub> reducing Vital Capacity deteriorating SpO<sub>2</sub>/ PaO<sub>2</sub>/ Vital Capacity improving/ stable O<sub>2</sub> needs reducing/ stable Pain score worse Pain controlled Continue regular reassessment and titration



Call 1213 for epidural/ block trouble shooting Re-site if necessary Contact ICU/ outreach
Consider Chest X-Ray
Consider NIV/ pasal high flow

Consider step down to non invasive pathway if sustained improvements



Figure 4: Rib fixation pathway

# Surgical Rib Fixation Pathway

Review by member of rib fracture fixation team.

Discussion & Decisions

- MDT may include: rib fracture fixation team, MTW consultant, anaesthetist, intensive care consultant, physiotherapist, occupational therapy & nursing staff.
- Decision for surgery made by 2 consultants.

Liaise with thoracic/ trauma surgeons if suspicion of large air leak or visceral injury.

If ipsilateral clavicle fractured, have low threshold for ORIF clavicle.

| Book | Half day theatre session. |
|---|---|
| Drugs | Give prophylactic LMWH ≥12 hours before planned surgery. |
| Equipment | MatrixRib fixation kit is sterile and available. |
| Imaging | 3D CT reconstruction thorax complete. |
| Blood results | FBC, renal profile (U&E & creatinine), clotting screen/ TEG. |
| Blood products | 2 units of packed red blood cells cross matched. |
| Anaesthetic team | <ol> <li>Insert thoracic epidural prior to anaesthetic induction if not already in situ OR ensure the dressings are distant to the operative site.</li> <li>Use standard single lumen endotracheal tube.</li> <li>Insert arterial line if anticipating NIV or inability to extubate.</li> </ol> |
| All theatre team | Position patient supine or laterally after discussion with surgeons |

Surgical team

Chest drains

 Plan surgical incision(s) by identifying fractures clinically or with ultrasound.
 If thoracic epidural not possible or contraindicated, insert paravertebral block/ catheter under direct vision at the end of the procedure.

3. Clean and debride original thoracostomy site to prevent infective complications.1. Replace any pre-existing chest drains prior to operative fixation through a new

thoracostomy

2. Insert a minimum of 1 chest drain per operated hemi-thorax at the end of the procedure and connect it to an underwater seal.

Mobile Chest X Ray at end of procedure in recovery or HDU to confirm drain position.

Post theatre destination

- 1. Aim to extubate at end of procedure. Arrange Major Trauma Ward/ Level 2 bed.
- 2. If intubated pre-op or significant respiratory compromise, to remain intubated and transfer back to ICU.
- 1. Give epidural levobupivacaine 0.125%/ fentanyl 2 mcg/ml mixture at 15 mls/hr.

Analgesia 2. Remove epidural 3-5 days after insertion (7 days maximum, if tunnelled, at discretion of anaesthetist & pain team).

3. Follow the invasive pathway



1. Regular ACBT and physiotherapy Rehabilitate 2. Sit up and ambulate ASAP. 1. Continue ACBT at home 4 hourly. Discharge planning 2. Wound review at 2 weeks.



Figure 5: Rib fracture tertiary referral form





# NORTH WEST LONDON TRAUMA NETWORK RIB FRACTURE TERTIARY REFERRAL FORM

| Referral details | | | | | |
|---|---|---|---|---|---|
| | Responsible Consultant: | | | | |
| | Contact telephone | | | | |
| Referring | (mobile): | | | | |
| clinician | Contact e-mail address: | | | | |
| | Hospital | | | | |
| | Ward | | | | |
| | Name: | | | | |
| | Date of birth: | | | | |
| Patient | NHS number: | | <i>,</i> | | |
| | Home address: | | | | |
| | General Practitioner: | | | | |
| Injury | | | | | |
| Mechanism: | | | | | |
| Rib fractures: | | | | | |
| Pneumothorax? Y | es No Haemo | othorax? Yes N | o Pulmonar | y contusion? Yes | No |
| Associated injurie | S: | | | | |
| Intomontions | | | | | |
| Interventions | V N Date | . Circumita d | / Deveio | tont oir look? Voo | NI - |
| Intercostal drain? | | of insertion:/ | / Persis | tent air leak? Yes | No |
| Imaging and findi | | | | | |
| | st (including 3D reconstructi | on rendered image | es) transferred by IEP: ` | Yes No | |
| Thoracic epidural | | | | | |
| Ventilation: | Self-ventilating | Non-ir | nvasive ventilation | Intubated | |
| FiO <sub>2</sub> | | AB | G results | | |
| Details of any oth | er treatment/surgery receive | <u>:d:</u> | | | |
| Pre-morbid state | | | | | |
| Co-morbidities: | | | | | |
| Previous thoracic | | | | | |
| cardiac/ thoracic | | | | | |
| surgery: | - I | | | | |
| , | | | | | l |



| | Imperial College Healthcare NHS Trust |
|-----------------------|---------------------------------------|
| Anticoagulant history | |
| including VTE | |
| prophylaxis: | |

Please e-mail referral to imperial.ribfracture@nhs.net



# 5) IMPLEMENTATION

| Training required for staff | ✓ Yes □ No |
|---|---|
| If yes, who will provide training: | Anaesthetic department: Epidurals and RA techniques |
| | Major Trauma Department: overall management |
| When will training be provided? | At induction of junior doctors, new consultants and regularly at nursing updates. |
| Date for implementation of guideline: | 1/3/2019 |

#### 6) MONITORING / AUDIT

| When will this guideline be audited? | Ongoing currently (clinical governance reference number 1850) |
|---|---|
| Who will be responsible for auditing this guideline? | Dr Alex Wickham, Consultant Anaesthetist<br>Mr Ian Sinha, Consultant Orthopaedic Surgeon |
| Are there any other specific recommendations for audit? | None |

# 7) REVIEW

| Frequency of review | Please indicate frequency of review: 3 years |
|---|---|
| | Person and post responsible for the review: Mr Ian Sinha, Consultant Orthopaedic Surgeon Dr Alex Wickham, Consultant Anaesthetist |

#### 8) REFERENCES

- 1. EAST Practice Management Guidelines Work Group. Pain management in Blunt Thoracic Trauma. *J Trauma* 2005; **59(5)**:1256-1267.
- 2. Battle C et al. Predicting outcomes after blunt chest wall trauma: development and external validation of a new prognostic model. *Crit Care* 2014, **18**:R98.
- 3. Witt C & Bulger E. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. *Trauma Surg Acute Care Open* 2017; **2**:1–7.
- 4. Galvagno SM Jr, Smith CE, Varon AJ, Hasenboehler EA, Sultan S, et al. Pain management for blunt thoracic trauma: a joint practice management guideline from the Eastern Association for the Surgery of Trauma and Trauma Anesthesiology Society. *J Trauma Acute Care Surg* 2016; **81**:936–51.
- 5. Jones KM, Reed RL, 2nd, Luchette FA. The ribs or not the ribs: which influences mortality? *Am J Surg*. 2011; **202(5)**:598Y604.
- 6. May L, Hillermann C & Patil S. Rib Fracture Management. BJA Education 2016; 16(1):26-32
- 7. Unsworth A, Curtis K & Asha SE. Treatments for blunt chest trauma and their impact on patient outcomes and health service delivery. *Scandinavian Journal of Trauma, Resuscitation and Emergency Medicine*, 2015; **23**:17
- 8. Butts C et al. Do simple beside lung function tests predict morbidity after rib fractures? *Am J Surg* 2017; **213(3)**:473-477.
- 9. Carver T, Milia D, Somberg C, Brasel K & Paul J. Vital capacity helps predict pulmonary complications after rib fractures. *J Trauma Acute Care Surg* 2015; **79(3)**:413-6.
- 10. Gordy S et al. The contribution of rib fractures to chronic pain and disability. Am J Surg 2014; 207(5): 659-62.
- 11. Royal College Of Anaesthetists. National Audit Project 3: Major Complications of Central Neuraxial Block in the United Kingdom. Report and Findings. January 2009. RCOA; London.



12. Carrier F, Turgeon A, Nicole P et al. Effect of epidural analgesia in patients with traumatic rib fractures: a systematic reviewand meta-analysis of randomized controlled trials. *Can J Anesth* 2009; **56**:230–242.



- 13. Jarvis AM, Cook CH, Lindsey DE, Reilley TE, Steinberg SM, Beery RM, Whitmill ML, Papadimos TJ, Stawicki SP. Comparison of epidural versus parenteral analgesia for traumatic rib fractures: A meta- analysis. *OPUS 12 Scientist* 2009; **3(3)**: 50-57.
- 14. Kunhabdulla NP, Agarwal A. Serratus Anterior Plane Block for Multiple Rib Fractures. *Pain Physician* 2014; 17: E651-662
- 15. Fu P, Weyker PD, Webb CAJ. Case Report of Serratus Plane Catheter for Pain Management in a Patient with Multiple Rib Fractures and an Inferior Scapular Fracture. *Anesth Analg* 2017;**8(6)**:132-135.
- 16. Marasco SF, Davies AR, Cooper J, Varma D, Bennett V, Nevill R, Lee G, Bailey M, Fitzgerald M. Prospective randomised controlled trial of operative rib fixation in traumatic flail chest. *J Am Coll Surg* 2013; **216(5)**:924-32.
- 17. Ahmed Z, Mohyuddin Z. Management of flail chest injury: internal fixation versus endotracheal intubation and ventilation. *J Thorac Cardiovasc Surg.* 1995; **110**:1676-80.
- 18. Tanaka H, Yukioka T, Yamaguti Y, et al. Surgical stabilization or internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. *J Trauma*. 2002; **52**:727–732.
- 19. Lafferty PM, Anavian J, Will RE, et al. Operative treatment of chest wall injuries: indications, technique, and outcomes. *J Bone Joint Surg Am* 2011; **93**:97–110.
- 20. Marasco SF, Davies AR, Cooper J, Varma D, Bennett V, Nevill R, Lee G, Bailey M & Fitzgerald M. Prospective Randomized Controlled Trial of Operative Rib Fixation in Traumatic Flail Chest. *J Am Coll Surg* 2013;**216**:924-932.
- 21. Bottlang M, Walleser S, Noll M, et al. Biomechanical rationale and evaluation of an implant system for rib fracture fixation. *European Journal of Trauma and Emergency Surgery* 2010; **36(5)**:417–426.
- 22. National Institute for Health and Care Excellence (NICE). *Interventional procedure guidance 361: Insertion of metal rib reinforcements to stabilise a flail chest wall.* 2010. NICE: London. Available from: <a href="https://www.nice.org.uk/guidance/ipg361">https://www.nice.org.uk/guidance/ipg361</a>
- 23. Adhikary S, Liu W, Fuller E, Cruz-Eng H and Chin K. The effect of erector spinae plane block on respiratory and analgesic outcomes in multiple rib fractures: a retrospective cohort study. *Anaesthesia* 2019; published online https://doi.org/10.1111/anae.14579
- 24. Todd S et al. A multidisciplinary clinical pathway decreases rib fracture—associated infectious morbidity and mortality in high-risk trauma patients. *Am. J Surg* 2006; **192**: 806–811.



# 9) **GUIDELINE DETAIL**

| Start Date: | 27 <sup>th</sup> August 2019 |
|---|---|
| Approval Dates | Anaesthetics and Major Trauma January 2015 Surgery, Cardiovascular and Cancer |
| | Major Trauma Board January 2015 |
| | <b>Drugs and therapeutics Committee</b> 26 <sup>th</sup> March 2019 (chair's action 2 <sup>nd</sup> April 2019 and 27 <sup>th</sup> August 2019) |
| Has all relevant legislation, | Please list ALL guidance considered: |
| national guidance, | |
| recommendations, alerts and | National Institute for Health and Care Excellence (NICE). |
| Trust action plans been | Interventional procedure guidance 361: Insertion of metal rib |
| considered, and included as appropriate in the development of this guideline? | reinforcements to stabilise a flail chest wall. 2010. NICE: London. |
| Have all relevant stakeholders | Please list all (name and role): |
| been included in the | Mr C Aylwin, Consultant trauma and vascular surgeon |
| development of this guideline? | Mr S Hettiaratchy, Consultant plastic surgeon |
| | Surg Commander M Khan, Consultant trauma surgeon |
| | Mr I Sinha, Consultant orthopaedic surgeon |
| | Dr S Qureshi, Consultant Anaesthetist |
| | Miss N Batrick, Consultant Emergency Physician & NWL Network lead |
| | Dr V Garnelo Rey, Consultant Intensivist & Trauma Lead |
| | Dr B Graham, Consultant Anaesthetist & Service Director |
| | Dr G Peck, Consultant Geriatrician |
| | St Mary's pain service: Dr J Illingworth, Dr A Knaggs, CNS A Fiamavle |
| | Dr B Bellew, Consultant Anaesthetist |
| | Mr K Bharkhada, Lead Pharmacist for Major Trauma and Pharmacy |
| | Miss N Marroney, Major Trauma Physiotherapist |
| | Mrs J Lockwood, Major Trauma Matron |
| | S H Jama, Senior Lead Pharmacist – Emergency, Acute and Elderly Medicine |
| | M Balic, Senior Lead Formulary Pharmacist and New Drugs Panel |
| Who will you be notifying of the | Secretary All clinical staff groups who are involved with the care of |
| existence of this guidance? | adult inpatients with rib fractures. |
| Related documents | Epidural Analgesia: Continuous Infusions Clinical Guidelines |
| | for Adult Patients |
| | Ketamine use for analgesia Guideline |
| | Pain management guidelines for adult patients with acute or chronic pain |
| | Analgesia Guideline for the Management of Acute and Chronic Pain for Adults with Renal Impairment |



| Author/further information | Name: Dr A Wickham, Mr I Sinha, Dr S Qureshi |
|---|---|
| | Title: Consultant Anaesthetist, Consultant Surgeon, Consultant |
| | Anaesthetist |
| | Division: Surgery, Cancer & Cardiovascular |
| | Site: St Mary's Hospital |
| | Telephone/Bleep: 26162 |
| | Trust email address: Alex.Wickham@nhs.net, |
| | Ian.Sinha1@nhs.net, Sabeena.Qureshi@nhs.net |

| Document review history | Next review due: 2 <sup>nd</sup> April 2022 |
|---|---|
| | Version 1: Major Trauma Board review July 2015 Version 2: DTC review and recommendations 26/3/19 Version 2.1: Update to CDU criteria |
| THIS GUIDELINE REPLACES: | Rib Fractures in Major Trauma: a guideline for management version 1, July 2015 |

# **10) INTRANET HOUSEKEEPING**

| Key words | Major Trauma, Rib Fracture, Epidural, Rib fixation |
|---|---|
| Which Division/Directorate category does this belong to? | Surgery, Cancer & Cardiovascular |
| Which specialty should this belong to when appearing on the Source? | Major Trauma |

**11) EQUALITY IMPACT OF GUIDELINE**Is this guideline anticipated to have any significant equality-related impact on patients, carers or staff? No **√**